CLINICAL TRIAL: NCT06822309
Title: Bilateral External Oblique Intercostal Plane Block Versus Patient Controlled Analgesia (PCA) in Post Operative Pain Management in Hepatectomy Surgery.
Brief Title: Bilateral External Oblique Intercostal Plane Block in Post Operative Pain Management in Hepatectomy
Acronym: EOI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sherif Alaa Embaby (Other)
Responsible Party: Sponsor-Investigator, Sherif Alaa Embaby, Consultant of Anaesthesia, ICU and pain management., Kasr El Aini Hospital
Organization: Kasr El Aini Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MS-189-2024
Record Dates: First submitted 2025-02-06; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Provide Post Hepatectomy Pain Control
Keywords: External Oblique Intercostal block; subcostal incision; hepatectomy; Patient control analgesia
MeSH Terms: interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- External Oblique Intercostal Plane block (Experimental): Patients in this group will receive External Oblique Intercostal plane block intraoperatively before the surgery.
  Interventions: Procedure: External Oblique Intercostal Plane Block
- Patient controlled analgesia (Active Comparator): Patient will be on patient control analgesia after the surgery.
  Interventions: Device: Patient controlled analgesia

INTERVENTIONS:
Procedure: External Oblique Intercostal Plane Block — The block is performed before skin incision by a specialized anesthetist. With the patient positioned in the supine position with their ipsilateral arm abducted, the skin was sterilized, using the high frequency linear probe (M-Turbo HF 38 transducer 13- 6 MHz) of Fujifilm Sonosite ultrasound is placed over the sixth rib medial to the anterior axillary line approximately in midclavicular line in a parasagittal orientation. A 20-guage needle is inserted in a cephalocaudal direction, and the external oblique intercostal plane was hydro dissected with saline. After hydro dissection, the needle is advanced 1 to 2 cm, and 20 mL of 0.25% bupivacaine (Sunny Pharmaceutical) with 4 mg dexamethasone as an additive was administered. The same procedure will be done at the other side (bilateral external oblique intercostal plane block).
  Arms: External Oblique Intercostal Plane block
Device: Patient controlled analgesia — Patients in group will receive intravenous patient controlled analgesia device 100 ml (Accuafuser 100 mL, basal rate 4 mL/hr., bolus 0.5 mL/time, and lock time 15 minutes) for postoperative pain management that will contain 30 mg morphine (loading dose0.1mg/kg) will be given by infusion over 10 minutes then accuafuser will be connected),8 mg dexamethasone and 8 mg ondansetron diluted in 100 ml saline.
  Arms: Patient controlled analgesia

SUMMARY:
The majority of cases undergoing hepatectomy suffer from inadequate postoperative analgesia. Therefore, multimodal analgesic techniques are required to relieve pain and discomfort such as intravenous, and epidural analgesia, and peripheral nerve blocks. Although epidural catheters are efficient to provide perioperative analgesia, in this type of surgery patients may be more susceptible to catheter related complications due to the alteration in coagulation parameters. That is why safer alternatives are sought for those patients. The use of patient-controlled analgesia (PCA) for postoperative pain management improves patients' quality of recovery. However, there are many concerns regarding the type of opioids used in PCA such as overdosing, underdosing, and the effect of the hepatectomy on the drug metabolism in those patients. External oblique intercostal plane block (EOI block) is a relatively novel block used in upper abdominal incisions especially subcostal laparotomy to provide intraoperative and postoperative analgesia.

This study aims to compare the efficacy of Bilateral External Oblique Intercostal Plain Block versus PCA in pain management and reduction of opioid use in hepatectomy surgery done by subcostal incision.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 65 Years.
* Both sexes.
* Patients will be scheduled for hepatectomy surgery.
* Body mass index (BMI) 18.5-30.0 /m 2 .

Exclusion Criteria:

* Extension of the surgical incision beyond coverage of T12 dermatome.
* Prolonged time of surgery > 5 hours.
* Hepatectomy surgery combined with another organ resection.
* Patients with hypersensitivity to local anesthetics.
* History of psychiatric problems.
* Recent history of analgesic drugs including opioid abuse or addiction.
* Coagulopathy (International normalized ratio [INR] > 1.4).
* Localized infection at the block site.
* Morbidly obese patients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
• Rescue morphine consumption in both groups. (Total consumption of morphine rescue shots in milligram in first 2r hours) | twenty four hours.

IPD SHARING:
Plan to Share IPD: Undecided
Once the study is over and published, all the data will be available.

REFERENCES:
- [Background] Cosarcan SK, Ercelen O. The analgesic contribution of external oblique intercostal block: Case reports of 3 different surgeries and 3 spectacular effects. Medicine (Baltimore). 2022 Sep 9;101(36):e30435. doi: 10.1097/MD.0000000000030435. PMID 36086688